CLINICAL TRIAL: NCT03951311
Title: Estimation of Metabolic Abnormalities,Lifestyle Behaviors and Diet Pattern in Adults With Heart Failure
Brief Title: Metabolic Abnormalities, Lifestyle and Diet Pattern in Heart Failure
Acronym: MALD-HF
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhijun Wu, Principal Investigator of department of cardiology, Ruijin Hospital
Other Study IDs: RJ-20172004
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Metabolic Disease
MeSH Terms: conditions — Heart Failure; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Fasting venous blood samples were drawn and transfused into vacuum tubes containing EDTA after admission. These samples were stored and further analyzed in the Central Laboratory of Ruijin Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic abnormalities (e.g., hypertension, diabetes mellitus, dyslipidemia, and obesity) and unhealthy lifestyle behaviors (e.g., smoking and drinking habits, sedentary behavior, sleep disorder and physical inactivity) and unhealthy diet (e.g., high sugar and high fat) are major risk factors for cardiovascular diseases mobility and mortality. The investigators sought to estimate the impact of metabolic abnormalities, lifestyle behavior and diet pattern on prognosis of heart failure. This study planned to consecutively enroll 1,500 participants with heart failure with reduced ejection fraction and heart failure with mid-range ejection fraction fulfilling the inclusion criteria. Each heart failure survivors will be followed up for 5 years. Information on metabolic diseases, lifestyle and diet pattern were obtained through standardized questionnaire. The major adverse cardiac events will be identified by reviewing pertinent medical records and discharge lists from the hospitals, or official death certificates collected at local death registration centers, or directly contacting participants' family. The Cox proportional hazard model will be used to assess the association between metabolic risk factors and lifestyle and diet habits and health outcomes in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged 14 years or older;
2. typical symptoms of heart failure according to the Framingham criteria;
3. left ventricular ejection fraction (LVEF) <50%, demonstrated by echocardiography or cardiac magnetic resonance, which include either patients with mid-range EF (HFmEF) or with reduced EF (HFrEF) with relevant structural and functional cardiac changes and/or elevated N-terminal pro-brain B-type natriuretic peptide (pro-BNP) (e.g., ≥400 pg/mL).

Exclusion Criteria:

1. age <14 years or ≥90 years;
2. pregnancy;
3. cancer with a life expectancy of less than one year;
4. participation in other trials;
5. endocarditis, pericardial diseases, or congenital heart diseases;
6. heart failure secondary to non-cardiac diseases (e.g., pulmonary heart disease, infection, infiltration, metabolic derangements, severe anemia, sepsis, and arteriovenous fistula);
7. lack of informed consent;
8. refusal of the drug treatment or intervention recommended by the guidelines.

Ages: 14 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients diagnosed with heart failure who had impaired cardiac function or abnormal cardiac structure with elevated blood BNP concentrations
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
a composite of cardiovascular mortality or hospitalization due to subjectively and objectively worsening HF | 5 years
  An independent committee of experts including three physicians reviews all the death certificates and medical records for adjudicating the death cases and all suspected CVD cases biennially from the index episode, via telephone contacting patients' family members or reviewing medical records and the Hospital Discharge Register data.

SECONDARY OUTCOMES:
cardiovascular mortality | 5 years
  sudden death or deaths due to CVD events
hospitalization due to worsening HF | 5 years
  the adjudicated hospitalizations due to subjectively and objectively worsening HF

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Wu, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Jin Y, Huang H, Zhou Q, Dong F, Lu L, Gao X, Wu Z. Prospective assessing metabolic abnormalities, lifestyle and dietary pattern in a Chinese population with heart failure: the MALD-HF study protocol. BMJ Open. 2022 May 2;12(5):e049225. doi: 10.1136/bmjopen-2021-049225. PMID 35501092